CLINICAL TRIAL: NCT05846529
Title: Assessment of Response Rate and Safety of Oral Thrombopoietin Receptor Agonist in Pediatric Chronic ITP in Assiut.
Brief Title: Safety of Oral Thrombopoietin Receptor Agonist in Pediatric Chronic ITP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salama Sayed Hassan, doctor, Assiut University
Other Study IDs: thrombopoietin agonist
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Thrombopoietin Receptor Agonist

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate the response rate and safety of oral thrombopoietin receptor agonist (Eltrombopag drug) used for children with chronic immune thrombocytopenia in patients attending Assiut university children's hospital.

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura (ITP) is an autoimmune disease characterized by decrease number of the platelets due to destruction of the platelets by antiplatelet antibodies. Also, platelet production can be reduced because the antiplatelet antibodies can also damage megakaryocytes . Its prevalence being approximately 8 per 100,000 children It is characterized by temporary or persistent reduction of the platelet number to less than 100 × 109/liter.

All new cases at diagnosis are defined as acute ITP. While, Persistent ITP is defined as ITP lasting between 3 and 12 months from diagnosis while chronic ITP is defined as the presence of ITP for more than one-year ITP Patients have an increased hazard of bleeding that may have no effect on patient's life or have life-threatening danger the goal of treatment in chronic ITP is to increase and then keep platelets in a sufficient number to prevent bleeding

. Meanwhile most life-threatening bleeding occurs with platelet number less than 30 × 109/liter.

New guideline recommend that treatment constricted on symptomatic patients with number lower than 30 × 109/liter (3,6) new Guidelines recommended that corticosteroids as first-line therapy and splenectomy considered as one of several second-line therapies. Other choices exist for ITP patients with insufficient response or who do not undergo to splenectomy including IVIg, IV anti-D, Rituximab, danazol, azathioprine, Vinca alkaloids and cyclophosphamide New consensus statements and guidelines recommend thrombopoietin-receptor (TPO-R) agonists as second and third line of treatment Eltrombopag consider the first oral, nonpeptide TPO-R agonist accepted for the treatment of chronic ITP in patients with insufficient response to at least one other therapy It rises platelet number by increase platelet production by binding to the transmembrane domain of the TPO-R. It does not compete with endogenous TPO in vitro and it enhance production and differentiation of BM progenitor cells in the megakaryocytic lineage

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 2 year and <18 years of age in both sex
* Confirmed diagnosis of chronic ITP
* all patient received oral thrombopoietin receptor agonist (Eltrombopag) for 6 months or more

Exclusion Criteria:

* age of the patient < 2years and >18 years
* secondary thrombocytopenia
* Concurrent or past malignant disease, including myeloproliferative disorder
* patient with platelet agglutination abnormality that prevents reliable measurement of platelet counts
* patient with bone marrow aplasia

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Infants and children between age of (2 year to <18 years old)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
response to oral thrombopoietin receptor agonist | baseline
  assess haematological response to oral thrombopoietin receptor agonist (Eltrombopag) therapy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuter DJ. The structure, function, and clinical use of the thrombopoietin receptor agonist avatrombopag. Blood Rev. 2022 May;53:100909. doi: 10.1016/j.blre.2021.100909. Epub 2021 Nov 16. PMID 34815110
- [Background] Jurczak W, Chojnowski K, Mayer J, Krawczyk K, Jamieson BD, Tian W, Allen LF. Phase 3 randomised study of avatrombopag, a novel thrombopoietin receptor agonist for the treatment of chronic immune thrombocytopenia. Br J Haematol. 2018 Nov;183(3):479-490. doi: 10.1111/bjh.15573. Epub 2018 Sep 7. PMID 30191972